CLINICAL TRIAL: NCT00841399
Title: Phase Ib Trial of HER2/Neu Peptide (E75) Vaccine in Breast Cancer Patients at Risk for Recurrence After Surgical and Medical Therapies
Brief Title: Safety and Efficacy Study of HER2/Neu (E75) Vaccine in Node-Positive Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: COL George Peoples, MD, FACS (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, COL George Peoples, MD, FACS, Chief, Surgical Oncology, Brooke Army Medical Center, Walter Reed Army Medical Center
Organization: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00-2005; WRAMC 20280 (Other: Walter Reed Army Med Center Institutional Review Board)
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- E75 + GM-CSF vaccine (Experimental): The dose escalation scheme is for three patients to receive each of the doses, 100, 500, and 1,000 mcg of peptide + 250 mcg GM-CSF each month for 6 months until the maximum tolerated dose is determined. Patients who receive the vaccine are HLA-A2+ and/or HLA-A3+. Responses to the vaccine are measured via immunologic assays.
  Interventions: Biological: E75 + GM-CSF vaccine
- Control/observation (No Intervention): HLA-A2- and HLA-A3- patients do not receive the E37 + GM-CSF vaccine, but are instead enrolled to the control arm for observation.

INTERVENTIONS:
Biological: E75 + GM-CSF vaccine — Dose escalation scheme involving three patients each receiving injection of 100, 500, or 1,000 mcg E75 + GM-CSF monthly for 6 months. HLA-A2 and HLA-A3 status determined. HLA-A2+ and HLA-A3+ patients receive the vaccine; HLA-A2- and HLA-A3- enrolled to the control arm.
  Arms: E75 + GM-CSF vaccine

SUMMARY:
The purposes of this study are the following:

1. To assess safety and document local and systemic toxicity to the peptide vaccine (E75)
2. To determine maximum tolerated dose (MTD) and optimal biologic dose (OBD) for the peptide vaccine
3. To evaluate the in vivo cellular immune response to the peptide vaccine
4. To evaluate time to recurrence in the vaccinated patients vs. matched controls

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy and second most common cause of cancer-specific death among women in the United States. Despite advances in the diagnosis and treatment of breast cancer, one third of the women who develop the disease will die of the disease, accounting for approximately 46,300 deaths/year. While good primary therapies are available to treat early stage breast cancer, there is a substantial failure rate to these therapies in more advanced disease.

Advances in the understanding of the immune response to cancer have lead to the genesis of immunotherapeutic approaches. Specifically, the development of anti-cancer vaccines holds promise as an adjuvant and preventive therapy for patients after both primary surgical and medical treatment for breast cancer, but who are at a high risk for recurrence. Patients with greater than four lymph nodes positive have an 87% chance of recurrence post standard surgical and medical therapies at 10 years. While patients with hormone receptor positive tumors have the option to undergo hormonal therapy, recurrence is especially high among estrogen receptor/progesterone receptor (ER/PR) negative patients. For these patients, currently there is no good treatment option after completion of primary therapy; close surveillance and watchful waiting is the standard.

It is this population of patients that a vaccine strategy to induce cellular immunity would target. We propose to vaccinate these patients with an immunogenic peptide from the HER2/neu protein. If successful, this vaccine strategy could be utilized as an adjuvant to currently accepted first line therapy in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. HER2/neu expressing tumor
2. HLA-A2+ and/or HLA-A3+ to receive the vaccine. HLA-A2- and/or HLA-A3- patients will be eligible to be included in the control group.
3. Immunologically intact with a good performance status
4. Identified as being high or intermediate risk for recurrence
5. Without evidence of disease
6. Completion of all standard first-line therapies (but may still be on hormonal therapy)

Exclusion Criteria:

1. Tumor does not express HER2/neu
2. Not HLA-A2+ and/or HLA-A3+
3. Anergic
4. Receiving immunosuppressive therapy
5. In poor health (Karnofsky <60%, ECOG >2 and Tbili >1.5 and creatinine>2)
6. Pregnant (beta HCG+)
7. Metastatic disease or have refused standard therapies
8. Patients enrolled in other experimental protocols may enroll to this study only with the permission of the other study PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2001-07; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoints are the safety and optimal dosing of the vaccine to induce an in vivo peptide-specific immune response. | Time period needed to determine the maximum tolerated and optimal biologic doses.

SECONDARY OUTCOMES:
The clinical endpoint is time to disease recurrence. | 30 days after each monthly vaccine, then per standard of care for breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: George E Peoples, MD, Principal Investigator — Cancer Vaccine Development Program
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Windber Medical Center, Windber, Pennsylvania

REFERENCES:
- [Background] Mittendorf EA, Storrer CE, Shriver CD, Ponniah S, Peoples GE. Investigating the combination of trastuzumab and HER2/neu peptide vaccines for the treatment of breast cancer. Ann Surg Oncol. 2006 Aug;13(8):1085-98. doi: 10.1245/ASO.2006.03.069. Epub 2006 Jul 24. PMID 16865596
- [Background] Dehqanzada ZA, Storrer CE, Hueman MT, Foley RJ, Harris KA, Jama YH, Kao TC, Shriver CD, Ponniah S, Peoples GE. Correlations between serum monocyte chemotactic protein-1 levels, clinical prognostic factors, and HER-2/neu vaccine-related immunity in breast cancer patients. Clin Cancer Res. 2006 Jan 15;12(2):478-86. doi: 10.1158/1078-0432.CCR-05-1425. PMID 16428490
- [Background] Woll MM, Fisher CM, Ryan GB, Gurney JM, Storrer CE, Ioannides CG, Shriver CD, Moul JW, McLeod DG, Ponniah S, Peoples GE. Direct measurement of peptide-specific CD8+ T cells using HLA-A2:Ig dimer for monitoring the in vivo immune response to a HER2/neu vaccine in breast and prostate cancer patients. J Clin Immunol. 2004 Jul;24(4):449-61. doi: 10.1023/B:JOCI.0000029117.10791.98. PMID 15163902
- [Result] Peoples GE, Gurney JM, Hueman MT, Woll MM, Ryan GB, Storrer CE, Fisher C, Shriver CD, Ioannides CG, Ponniah S. Clinical trial results of a HER2/neu (E75) vaccine to prevent recurrence in high-risk breast cancer patients. J Clin Oncol. 2005 Oct 20;23(30):7536-45. doi: 10.1200/JCO.2005.03.047. Epub 2005 Sep 12. PMID 16157940
- [Result] Mittendorf EA, Gurney JM, Storrer CE, Shriver CD, Ponniah S, Peoples GE. Vaccination with a HER2/neu peptide induces intra- and inter-antigenic epitope spreading in patients with early stage breast cancer. Surgery. 2006 Mar;139(3):407-18. doi: 10.1016/j.surg.2005.06.059. PMID 16546506
- [Result] Hueman MT, Stojadinovic A, Storrer CE, Dehqanzada ZA, Gurney JM, Shriver CD, Ponniah S, Peoples GE. Analysis of naive and memory CD4 and CD8 T cell populations in breast cancer patients receiving a HER2/neu peptide (E75) and GM-CSF vaccine. Cancer Immunol Immunother. 2007 Feb;56(2):135-46. doi: 10.1007/s00262-006-0188-9. Epub 2006 Jun 17. PMID 16783576
- [Result] Dehqanzada ZA, Storrer CE, Hueman MT, Foley RJ, Harris KA, Jama YH, Shriver CD, Ponniah S, Peoples GE. Assessing serum cytokine profiles in breast cancer patients receiving a HER2/neu vaccine using Luminex technology. Oncol Rep. 2007 Mar;17(3):687-94. PMID 17273752
- [Result] Stojadinovic A, Mittendorf EA, Holmes JP, Amin A, Hueman MT, Ponniah S, Peoples GE. Quantification and phenotypic characterization of circulating tumor cells for monitoring response to a preventive HER2/neu vaccine-based immunotherapy for breast cancer: a pilot study. Ann Surg Oncol. 2007 Dec;14(12):3359-68. doi: 10.1245/s10434-007-9538-x. Epub 2007 Sep 29. PMID 17906897
- [Result] Peoples GE, Holmes JP, Hueman MT, Mittendorf EA, Amin A, Khoo S, Dehqanzada ZA, Gurney JM, Woll MM, Ryan GB, Storrer CE, Craig D, Ioannides CG, Ponniah S. Combined clinical trial results of a HER2/neu (E75) vaccine for the prevention of recurrence in high-risk breast cancer patients: U.S. Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Clin Cancer Res. 2008 Feb 1;14(3):797-803. doi: 10.1158/1078-0432.CCR-07-1448. PMID 18245541
- [Result] Amin A, Benavides LC, Holmes JP, Gates JD, Carmichael MG, Hueman MT, Mittendorf EA, Storrer CE, Jama YH, Craig D, Stojadinovic A, Ponniah S, Peoples GE. Assessment of immunologic response and recurrence patterns among patients with clinical recurrence after vaccination with a preventive HER2/neu peptide vaccine: from US Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Cancer Immunol Immunother. 2008 Dec;57(12):1817-25. doi: 10.1007/s00262-008-0509-2. Epub 2008 Apr 8. PMID 18392824
- [Result] Mittendorf EA, Holmes JP, Ponniah S, Peoples GE. The E75 HER2/neu peptide vaccine. Cancer Immunol Immunother. 2008 Oct;57(10):1511-21. doi: 10.1007/s00262-008-0540-3. Epub 2008 Jun 7. PMID 18536917
- [Result] Holmes JP, Gates JD, Benavides LC, Hueman MT, Carmichael MG, Patil R, Craig D, Mittendorf EA, Stojadinovic A, Ponniah S, Peoples GE. Optimal dose and schedule of an HER-2/neu (E75) peptide vaccine to prevent breast cancer recurrence: from US Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Cancer. 2008 Oct 1;113(7):1666-75. doi: 10.1002/cncr.23772. PMID 18726994
- [Result] Holmes JP, Clifton GT, Patil R, Benavides LC, Gates JD, Stojadinovic A, Mittendorf EA, Ponniah S, Peoples GE. Use of booster inoculations to sustain the clinical effect of an adjuvant breast cancer vaccine: from US Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Cancer. 2011 Feb 1;117(3):463-71. doi: 10.1002/cncr.25586. Epub 2010 Sep 15. PMID 20845479
- [Result] Patil R, Clifton GT, Holmes JP, Amin A, Carmichael MG, Gates JD, Benavides LH, Hueman MT, Ponniah S, Peoples GE. Clinical and immunologic responses of HLA-A3+ breast cancer patients vaccinated with the HER2/neu-derived peptide vaccine, E75, in a phase I/II clinical trial. J Am Coll Surg. 2010 Feb;210(2):140-7. doi: 10.1016/j.jamcollsurg.2009.10.022. Epub 2009 Dec 22. PMID 20113933
- [Result] Mittendorf EA, Clifton GT, Holmes JP, Clive KS, Patil R, Benavides LC, Gates JD, Sears AK, Stojadinovic A, Ponniah S, Peoples GE. Clinical trial results of the HER-2/neu (E75) vaccine to prevent breast cancer recurrence in high-risk patients: from US Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Cancer. 2012 May 15;118(10):2594-602. doi: 10.1002/cncr.26574. Epub 2011 Oct 11. PMID 21989902
- [Result] Benavides LC, Sears AK, Gates JD, Clifton GT, Clive KS, Carmichael MG, Holmes JP, Mittendorf EA, Ponniah S, Peoples GE. Comparison of different HER2/neu vaccines in adjuvant breast cancer trials: implications for dosing of peptide vaccines. Expert Rev Vaccines. 2011 Feb;10(2):201-10. doi: 10.1586/erv.10.167. PMID 21332269
- [Result] Benavides LC, Gates JD, Carmichael MG, Patil R, Holmes JP, Hueman MT, Mittendorf EA, Craig D, Stojadinovic A, Ponniah S, Peoples GE. The impact of HER2/neu expression level on response to the E75 vaccine: from U.S. Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Clin Cancer Res. 2009 Apr 15;15(8):2895-904. doi: 10.1158/1078-0432.CCR-08-1126. Epub 2009 Apr 7. PMID 19351776
- [Result] Hueman MT, Stojadinovic A, Storrer CE, Foley RJ, Gurney JM, Shriver CD, Ponniah S, Peoples GE. Levels of circulating regulatory CD4+CD25+ T cells are decreased in breast cancer patients after vaccination with a HER2/neu peptide (E75) and GM-CSF vaccine. Breast Cancer Res Treat. 2006 Jul;98(1):17-29. doi: 10.1007/s10549-005-9108-5. Epub 2006 Jun 7. PMID 16758122
- [Derived] Mittendorf EA, Clifton GT, Holmes JP, Schneble E, van Echo D, Ponniah S, Peoples GE. Final report of the phase I/II clinical trial of the E75 (nelipepimut-S) vaccine with booster inoculations to prevent disease recurrence in high-risk breast cancer patients. Ann Oncol. 2014 Sep;25(9):1735-1742. doi: 10.1093/annonc/mdu211. Epub 2014 Jun 6. PMID 24907636